CLINICAL TRIAL: NCT04048460
Title: Assessment of e-Audiology for Providing Clinical Services and Support for Age-related Hearing Loss: A Pilot Study
Brief Title: Assessment of e-Audiology for Providing Clinical Services and Support
Acronym: eAudiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Victoria Sanchez (Williams), Assistant Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00041124
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Hearing Loss, Age-Related; Presbycusis, Bilateral; Hearing Disability
Keywords: telehealth; eAudiology; accessibility; Age-related hearing loss
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eAudiology (Experimental): Participants will receive bilateral, behind-the-ear hearing aids as part of this study. The intervention will involve e-Audiology sessions following the initial hearing aid fitting and orientation. E-Audiology sessions will consist of hearing aid follow-up programming, troubleshooting, HAT assistance, and general help with hearing devices. E-Audiology sessions will take place over the course of approximately 6 weeks.
  Interventions: Device: Delivery of hearing healthcare through eAudiology application

INTERVENTIONS:
Device: Delivery of hearing healthcare through eAudiology application — Participants will receive bilateral, behind-the-ear hearing aids as part of this study. The intervention will involve e-Audiology sessions following the initial hearing aid fitting and orientation. E-Audiology sessions will consist of hearing aid follow-up programming, troubleshooting, HAT assistance, and general help with hearing devices. E-Audiology sessions will take place over the course of approximately 6 weeks.

SUMMARY:
Technological advances in hearing aids and telecommunications, including the widespread availability of telehealth (referred to in this proposal as "e-Audiology") applications, have the potential to expand both access and affordability of hearing aids for those with age-related hearing loss (ARHL). E-Audiology is used by clinicians in a variety of settings, including private practice, university clinics, and the Veterans Administration. The American Speech-Language-Hearing Association recently updated the Scope of Practice guidelines for audiology to include telehealth as "an alternative method of service delivery that en-compasses both diagnostics and intervention services.", including all aspects of hearing aid selection, fitting, and follow-up counseling and rehabilitation. However, given the paucity of evidence of comparative efficacy between office-based service delivery and e-Audiology in real-world settings, patients and relevant stakeholders are faced with a major decisional dilemma when determining which mode of service delivery would be optimal for addressing the needs, preferences, and lifestyles of those with ARHL. Thus, the purpose of this study is to determine the benefits, drawbacks, and patient satisfaction associated with e-Audiology delivery of hearing aid fitting, services, and supports for older adults with mild to moderate ARHL. We plan to use data collected in this pilot study for a future R01 submission to the NIH.

DETAILED DESCRIPTION:
Hearing loss is a chronic disability and a major public health concern. As the U.S. population ages, hearing loss prevalence rates are expected to nearly double by 2060 (Goman, Reed et al. 2017). Given this projection and the negative, costly impacts of untreated hearing loss on health outcomes, there is a national emphasis on increasing access and affordability of hearing healthcare (HHC) (President's Council of Advisors on Science and Technology 2015, National Academies of Sciences 2016). Two significant factors hinder the achievement of successful HHC outcomes: First, US adults face structural barriers to accessing HHC including high cost, and limited, inflexible points of entry into the system (National Academies of Sciences 2016). Second, hearing aids are often the sole intervention offered. While hearing aids improve speech understanding in quiet, difficulties understanding speech in challenging listening environments remain. Many of these difficulties can be addressed by including hearing assistive technology [HAT] options in the intervention plan. Unfortunately, hearing aid uptake is low for adults with hearing loss, and HAT usage is reported among only a fraction of those who use hearing aids (Southall, Gagné et al. 2009, Hartley, Rochtchina et al. 2010, Chien and Lin 2012, Bainbridge and Ramachandran 2014). Technological advances in hearing aids and telecommunications, including the widespread availability of "e-Audiology" applications, have the potential to expand both access and affordability of HHC by allowing for greater flexibility, lower costs, and personalized intervention plans that take into account the listening and lifestyle needs of the individual. There is a lack of evidence, however, as to how e-Audiology and patient acceptance for e-Audiology impact HHC outcomes. There is an urgent need to understand the efficacy of accessible, patient-centered, and comprehensive HHC alternative delivery models, like e-Audiology, without which the critical public health problem of untreated hearing loss in adults will likely worsen.

With the long-term goal of enhancing decision-making by patients and providers and improving outcomes, the pilot data collected in this proposal will be used for an upcoming R01 submission which will be responsive to the NIDCD's call for research comparing different HHC delivery models and the utilization of new technologies to improve care. The overall objectives of this work are twofold. First, we will evaluate outcomes from an e-Audiology service delivery model. Second, we will determine the impact of patient preferences for delivery model on outcomes. The rationale of the proposed study is that the results will enhance the evidence-base for the use of e-Audiology as a mechanism for increasing HHC access for diverse adult populations. Results obtained will be submitted as pilot data in an upcoming R01 grant application.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Community-dwelling
* Can speak and read English fluently, assessed by self-report
* Mild to severe sloping hearing loss, as determined by a 4-frequency pure-tone average (0.5 to 4.0 kHz) of > 30 dB HL in the better ear and no greater than 90 dB at any frequency
* Cognitively intact, as determined by a Mini Mental State Exam (MMSE) score of 23 or greater
* Regular access to computer, tablet, or "smart device" capable of delivering the e-Audiology platform

Exclusion Criteria:

* Bilateral conductive hearing loss, defined as a > 10 dB air-bone gap at 2 or more frequencies
* Corrected vision no worse than 20/63, assessed by the MN Read Acuity vision screening
* Unwillingness to use hearing aids on a daily basis, determined by self-report

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Auditory Rehabilitation and Clinical Trials Laboratory at the University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- eAudiology: Participants received bilateral, behind-the-ear hearing aids as part of this study. The intervention involved e-Audiology sessions following the initial hearing aid fitting and orientation. E-Audiology sessions consisted of hearing aid follow-up programming, troubleshooting, HAT assistance, and general help with hearing devices. E-Audiology sessions took place over the course of approximately 6 weeks from baseline.
Period: Overall Study
Arm/Group | eAudiology
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- eAudiology: Participants received bilateral, behind-the-ear hearing aids as part of this study. The intervention will involved e-Audiology sessions following the initial hearing aid fitting and orientation. E-Audiology sessions will consisted of hearing aid follow-up programming, troubleshooting, HAT assistance, and general help with hearing devices. E-Audiology sessions took place over the course of approximately 6 weeks from baseline.
Arm/Group | eAudiology
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Unaided Quick Speech In Noise Test (QuickSIN) [Mean (Standard Deviation); unit: Decibels] — Participants repeat sentences presented at six signal-to-noise ratios (SNRs) and the 'SNR loss' is computed. The SNR loss is the dB SNR relative to the SNR required for normal hearing individuals to repeat back 50% of the key words correctly.
  Higher scores on the signal to noise ratio loss scale indicates more difficulty with hearing speech-in-noise compared to normal hearing peers. The range of performance is from 2-dB SNR to 24-dB SNR. Scores are reported as the average SNR loss across all participants at baseline.
  Decibels | 7.75 (5.75)
Hearing Handicap Inventory for the Elderly Screening (HHIE-S) [Mean (Standard Deviation); unit: Scores on a scale] — The Hearing Handicap Inventory for the Elderly Screening (HHIE-S) (Ventry and Weinstein 1982, Newman and Weinstein 1988) will be used to measure self-reported hearing difficulties.
  The Hearing Handicap Inventory scale is reported as an average across all participants and has a minimum value of 0 and a maximum value of 40. Higher scores indicate more perceived social and emotional difficulty due to an individuals hearing loss.
  Scores on a scale | 9.5 (2.72)
Telehealth Acceptance Questionnaire (TAQ) [Mean (Standard Deviation); unit: mm] — Telehealth Acceptance Questionnaire (TAQ; Wade, 2012). The TAQ is based on the Technology Acceptance Model, and will be used to assess participants' attitudes about telehealth as well as their beliefs regarding self-efficacy for telehealth use. The TAQ uses a visual analog scale and the units range from 0 mm (lowest acceptance of telehealth) to 100 mm (higher acceptance of telehealth). The scores are reported as an average across all participants.
  mm | 8.29 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Hearing Handicap Inventory for the Elderly Screening Version (HHIE-S)
Description: The Hearing Handicap Inventory for the Elderly Screening (HHIE-S) (Ventry and Weinstein 1982, Newman and Weinstein 1988) will be used to measure self-reported hearing difficulties.
  The Hearing Handicap Inventory scale is reported as an average across all participants and has a minimum value of 0 and a maximum value of 40. Higher scores indicate more perceived social and emotional difficulty due to an individuals hearing loss.
  Change in HHIE scores were calculated based on the change from baseline to 6 weeks-post intervention.
Time Frame: 6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | eAudiology
Number analyzed (Participants) | 10
scores on a scale | 3.2 (3.68)

2. Secondary Outcome: Change From Baseline on the Quick Speech-in-Noise (QuickSIN) Test
Description: Participants repeat sentences presented at six signal-to-noise ratios (SNRs) and the 'SNR loss' is computed. The SNR loss is the dB SNR relative to the SNR required for normal hearing individuals to repeat back 50% of the key words correctly.
  Higher scores on the signal to noise ratio loss scale indicates more difficulty with hearing speech-in-noise compared to normal hearing peers. The range of performance is from 2-dB SNR to 24-dB SNR. Scores are reported as the average SNR loss across all participants. The change in SNR loss was calculated based on the change in average score from baseline to 6-weeks post-intervention.
Time Frame: 6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | eAudiology
Number analyzed (Participants) | 10
Decibels | 5.0 (4.41)

3. Secondary Outcome: Change From Baseline on the Telehealth Acceptance Questionnaire (TAQ)
Description: Telehealth Acceptance Questionnaire (TAQ; Wade, 2012). The TAQ is based on the Technology Acceptance Model, and will be used to assess participants' attitudes about telehealth as well as their beliefs regarding self-efficacy for telehealth use. The TAQ uses a visual analog scale and the units range from 0 mm (lowest acceptance of telehealth) to 100 mm (higher acceptance of telehealth). The scores are reported as an average across all participants. Change from baseline was calculated based on the change in average score from baseline to 6-weeks post-intervention.
Time Frame: 6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | eAudiology
Number analyzed (Participants) | 10
mm | 8.79 (1.49)

4. Secondary Outcome: International Outcome Inventory for Hearing Aids (IOI-HA)
Description: The IOI-HA will be used to determine specific hearing aid benefits perceived by the participants following a sustained period of use. This a post-intervention measurement only as questions are specific to the intervention adopted.
  The International Outcome Inventory scale ranges from 7 to 35. A higher score would indicate more perceived benefit from hearing aids.
Time Frame: 6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eAudiology
Number analyzed (Participants) | 10
units on a scale | 31.9 (2.60)

ADVERSE EVENTS:
Time Frame: Non-serious/other adverse events were assessed from enrollment (signed consent) to end of study (final study assessment). The total duration of time in the study for each participant was an average of 6 weeks. Follow-up visits took place at regularly-scheduled, 2-week intervals following the baseline visit over the course of 6 weeks. Adverse event data was collected over this time period for each participant.
Description: Potential risks to participants in this study are minimal. There is a slight risk of boredom, anxiety, or fatigue associated with the questionnaires, hearing testing, hearing aid fitting, and/or follow-up hearing aid e-Audiology sessions. All test measures in this study are used routinely in clinical practice by audiologists for assessing hearing outcomes of clinical and research participants.
  Due to the nature of the study, all-cause mortality and serious adverse events were not assessed.
Arm/Group | eAudiology
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT04048460/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT04048460/ICF_001.pdf